CLINICAL TRIAL: NCT01562613
Title: Stroke Estimation (According to Framingham Profile ParameterS) in Patients Under medicAtion Due to Essential Hypertension. (NASA)
Brief Title: A Blood Pressure Regulation and Stroke Risk Evaluation Study in Hypertensive Patients Treated With Eprosartan
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P13-165
Record Dates: First submitted 2012-03-16; First posted 2012-03-26 (Estimated); Results first posted 2014-07-30 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension; Stroke
Keywords: Stroke; Hypertension
MeSH Terms: conditions — Hypertension; Stroke

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypertensive patients: All eligible hypertensive patients treated with eprosartan

SUMMARY:
The primary objective of the study is to evaluate the proportion of hypertensive patients who achieve regulation of their blood pressure (BP) levels according to the European Society of Cardiology / European School of Haematology (ESC/ESH) Guidelines, after treatment with eprosartan for 6 months under standard medical practice conditions. The absolute change in Systolic blood pressure from baseline will also be calculated.

This study also aims in the evaluation of Framingham stroke risk profile score of patients treated with eprosartan under standard clinical practice conditions during the observation period. Besides the primary and the secondary objective of the study, the assessment of the percentage of patients who experienced Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Drug Reactions (ADRs), Serious Adverse Drug Reactions (SADRs) (overall and per observed event) and the percentage of patients who discontinued treatment prematurely before the advent of the 6-month observation period due to toxicity to the study medication constitutes another important objective that is related to the safety of the treatment.

DETAILED DESCRIPTION:
This is an open, non-interventional, non-comparative study. Therefore, there is no control group, randomization, or blinding involved. The target subject population is hypertensive patients who are being treated with eprosartan under standard clinical conditions and the locally approved Summary of Product Characteristics (SmPCs). Treatment selection is independent of the study conduct according to the local requirements of the Health Authorities for the definition of non-interventional studies being conducted in Greece. Therefore, the inclusion/exclusion criteria of this study follow the clinical decision of the participating physician, when prescribing the study medication(s) under standard clinical practice. The study plans to enroll 600 patients from 100 participating centers (hospitals and private physicians). This number includes an additional 25% cushion compared to the required sample size to ensure that sufficient data is collected for the subsequent statistical analysis. The study has been designed to be non-interventional and subsequently follows the per center standard practice of treatment, medical care and visits. As a result a rigid visit schedule could not be imposed. However, when taking into account the overall local standard practice, an overview of the visit schedule is indicated per subject:

* A baseline visit at the beginning of the 6-month observation period where the investigator will check the eligibility of the subject and will record the baseline data provided that the subject is eligible and has given the signed and dated informed consent.
* A final visit at the end of the 6-month treatment period (also observation period), and
* At least one interim visit (according to the standard clinical practice, within baseline and final visit)

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age greater or equal to 18 years)
2. Hypertensive patients, with a sitting Systolic Blood Pressure above 140 mmHg or 130 mmHg in diabetics and high/very high risk patients, according to ESC/ESH Guidelines
3. Patients being prescribed eprosartan under the terms and conditions of the local label and administered according to standard medical practice
4. Patients with at least one of the following conditions:

   * Newly diagnosed hypertension,
   * Inability to tolerate other antihypertensive medications, or
   * Lack of response to current antihypertensive medication(s)

Exclusion Criteria:

1. Any contraindication to eprosartan or the excipients (according to the local label)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with eprosartan according to routine medical practice from hospitals and private physicians.
Sampling Method: Non-Probability Sample
Enrollment: 533 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Daskalaki, MD, Study Director — Abbott
Locations (84):
- Greece (84):
  - Site Reference ID/Investigator# 62499, Agrinio
  - Site Reference ID/Investigator# 62500, Agrinio
  - Site Reference ID/Investigator# 62577, Alimos
  - Site Reference ID/Investigator# 62386, Athens
  - Site Reference ID/Investigator# 62398, Athens
  - Site Reference ID/Investigator# 62389, Athens
  - Site Reference ID/Investigator# 62384, Athens
  - Site Reference ID/Investigator# 62392, Chalandri
  - Site Reference ID/Investigator# 62395, Chalandri
  - Site Reference ID/Investigator# 62391, Chalandri
  - Site Reference ID/Investigator# 62633, Chalcis
  - Site Reference ID/Investigator# 62629, Chalcis
  - Site Reference ID/Investigator# 62507, Chania
  - Site Reference ID/Investigator# 62508, Chania
  - Site Reference ID/Investigator# 62511, Chania
  - Site Reference ID/Investigator# 62588, Chania
  - Site Reference ID/Investigator# 62484, Drama
  - Site Reference ID/Investigator# 62518, Eleftherio, Thessaloniki
  - Site Reference ID/Investigator# 62512, Euosmos, Thessaloniki
  - Site Reference ID/Investigator# 62390, Galatsi
  - Site Reference ID/Investigator# 62584, Glyfada
  - Site Reference ID/Investigator# 62586, Glyfada
  - Site Reference ID/Investigator# 62589, Heraklion
  - Site Reference ID/Investigator# 62591, Heraklion
  - Site Reference ID/Investigator# 62505, Heraklion
  - Site Reference ID/Investigator# 62593, Heraklion
  - Site Reference ID/Investigator# 62587, Heraklion
  - Site Reference ID/Investigator# 62503, Ioannina
  - Site Reference ID/Investigator# 62497, Ioannina
  - Site Reference ID/Investigator# 62493, Ioannina
  - Site Reference ID/Investigator# 62487, Kalamata
  - Site Reference ID/Investigator# 62580, Kallithea
  - Site Reference ID/Investigator# 62645, Kavala
  - Site Reference ID/Investigator# 62644, Kavala
  - Site Reference ID/Investigator# 62483, Komotini
  - Site Reference ID/Investigator# 62642, Komotini
  - Site Reference ID/Investigator# 62575, Korydallos
  - Site Reference ID/Investigator# 62631, Lamia
  - Site Reference ID/Investigator# 62635, Lamia
  - Site Reference ID/Investigator# 62626, Larissa
  - Site Reference ID/Investigator# 62638, Larissa
  - Site Reference ID/Investigator# 62628, Larissa
  - Site Reference ID/Investigator# 62637, Larissa
  - Site Reference ID/Investigator# 62574, Megara
  - Site Reference ID/Investigator# 62630, N. Ionia Volou
  - Site Reference ID/Investigator# 62397, Néa Erythraía
  - Site Reference ID/Investigator# 62385, Néa Filadélfeia
  - Site Reference ID/Investigator# 62399, Néa Smýrni
  - Site Reference ID/Investigator# 62582, Nikaia
  - Site Reference ID/Investigator# 62585, P. Faliro
  - Site Reference ID/Investigator# 62393, Paianía
  - Site Reference ID/Investigator# 62394, Pallini
  - Site Reference ID/Investigator# 62522, Panórama
  - Site Reference ID/Investigator# 62501, Pátrai
  - Site Reference ID/Investigator# 62502, Pátrai
  - Site Reference ID/Investigator# 62492, Pátrai
  - Site Reference ID/Investigator# 62401, Peristeri
  - Site Reference ID/Investigator# 62402, Peristeri
  - Site Reference ID/Investigator# 62578, Peristeri
  - Site Reference ID/Investigator# 62388, Peuki
  - Site Reference ID/Investigator# 62396, Peuki
  - Site Reference ID/Investigator# 62579, Piraeus
  - Site Reference ID/Investigator# 62520, Polykastro
  - Site Reference ID/Investigator# 62495, Pýrgos
  - Site Reference ID/Investigator# 62496, Pýrgos
  - Site Reference ID/Investigator# 62510, Rhodes
  - Site Reference ID/Investigator# 62590, Rhodes
  - Site Reference ID/Investigator# 62592, Rhodes
  - Site Reference ID/Investigator# 62640, Sappes Komotinis
  - Site Reference ID/Investigator# 62641, Serres
  - Site Reference ID/Investigator# 62513, Sykiés
  - Site Reference ID/Investigator# 62509, Thermi, Thessaloniki
  - Site Reference ID/Investigator# 62514, Thessaloniki
  - Site Reference ID/Investigator# 62517, Thessaloniki
  - Site Reference ID/Investigator# 62516, Thessaloniki
  - Site Reference ID/Investigator# 62521, Thessaloniki
  - Site Reference ID/Investigator# 62523, Thessaloniki
  - Site Reference ID/Investigator# 62506, Véria
  - Site Reference ID/Investigator# 62627, Volos
  - Site Reference ID/Investigator# 62634, Volos
  - Site Reference ID/Investigator# 62486, Vraxnaiika
  - Site Reference ID/Investigator# 62387, Výronas
  - Site Reference ID/Investigator# 62485, Xánthi
  - Site Reference ID/Investigator# 62488, Xánthi

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypertensive Patients
Started | 533
Completed | 529
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 533
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 276
  Male | 257
Region of Enrollment [Number; unit: participants]
  Greece | 533

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Hypertensive Patients Who Achieve Regulated BP Levels According to the ESC/ESH Guidelines, After They Have Been Treated With Eprosartan for 6 Months Under Standard Daily Medical Practice Conditions.
Description: The percentage of hypertensive patients who achieve regulated BP levels according to the ESC/ESH (European Society of Cardiology/European Society of Hypertension) Guidelines, after they have been treated with eprosartan for 6 months under standard daily medical practice conditions.
  Rate of responders (%) who reach the ESH/ESC Guidelines BP levels of <140 mmHg/90 mmHg [systolic BP (SBP)/diastolic BP (DBP)] for the general population of hypertensive patients OR of <130 mmHg/80 mmHg in case of diabetics and high or very high risk patients such as those with associated clinical conditions [stroke, myocardial infarction, coronary artery disease (CAD)]
Time Frame: Baseline up to 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 529
Percentage of participants | 62.8 [58.6 to 66.9]

2. Primary Outcome: The Absolute Change in Systolic Blood Pressure From Baseline
Description: The absolute change in systolic Blood Pressure from baseline
Time Frame: Baseline up to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 529
mmHg | -31.1 (11.9)

3. Secondary Outcome: Change in Framingham Stroke Risk Profile Scores of the Participating Patients
Description: The Framingham Stroke Risk Profile assesses the Probability of Stroke Within 10 Years separately for a) Women Aged 55-84 Years and Free of Previous Stroke AND b) for Men Aged 55-85 Years and Free of Previous Stroke.
  First the Framingham Stroke Risk Profile Score is calculated as the sum of points obtained from each of the following factors: age, treated or untreated SBP, presence of diabetes, cigarette smoking, cardiovascular disease, atrial fibrillation, hypertension, and left ventricular hypertrophy according to the gender-specific tables provided by D'Agostino et al (Stroke 1994: 40-43). Subsequently the total score obtained yields the 10-year probability of stroke from gender-specific tables provided in D'Agostino et al.
  The score can range from 0-38 (according to the scales of D' Agostino et al) with higher scores yielding increased 10-year probability of stroke.
Time Frame: Baseline up to 6 months
Population: Excluded from Framingham calculation were patients with either
  1. a history of cerebrovascular accident
  2. any of the parameters missing for the calculation of the Framingham
  3. age <54 years or > 84 years for females & <54 or > 85 years for males
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Hypertensive Patients
Number analyzed (Participants) | 370
score on a scale
  Baseline | 14 (1.7) [4 to 29]
  6 months | 11 [3 to 27]

ADVERSE EVENTS:
Arm/Group | Hypertensive Patients
Serious Adverse Events (participants affected / at risk) | 0/533
Other Adverse Events (participants affected / at risk) | 7/533
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypertensive Patients (N=533)
Gastroenteritis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Dizziness (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No important limitations apply. Missing data and drop-out rate was very low; but some factors required for patient CV (cardiovascular) risk classification were unknown and may have resulted in CV risk underestimation in a limited number of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days